CLINICAL TRIAL: NCT04652674
Title: Impact of Postoperative Telemedicine Visit vs In-person Visit on Patient Satisfaction During the COVID-19 Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Karen Zaghiyan, Associate Professor of Surgery, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00000944
Record Dates: First submitted 2020-12-02; First posted 2020-12-03 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Covid19; Satisfaction, Patient; Telemedicine
Keywords: Covid19; Patient satisfaction; Telemedicine
MeSH Terms: conditions — COVID-19; Patient Satisfaction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): Patients who will undergo telemedicine visit approximately 1 week postoperatively, then an in-person clinic visit approximately 4 weeks postoperatively
  Interventions: Behavioral: Telemedicine visit
- Group II (Active Comparator): Patients who will undergo in-person clinic visit approximately 1 week postoperatively, then a telemedicine visit approximately 4 weeks postoperatively
  Interventions: Behavioral: In-person postoperative visit

INTERVENTIONS:
Behavioral: Telemedicine visit — A postoperative visit with the patient's surgeon conducted remotely via audio/video smartphone app
  Other Names: Remote audio/video visit, telehealth visit
  Arms: Group I
Behavioral: In-person postoperative visit — A standard-of-care in-person postoperatively visit with the patient's surgeon
  Arms: Group II

SUMMARY:
The purpose of this clinical study is to evaluate whether remote video/audio postoperative visits (telemedicine visits) affects patient satisfaction compared to in-person visits during the COVID-19 pandemic. If the primary objective of the study is achieved, it would allow better understanding of how telemedicine can be integrated into modern surgical practice to take care of postoperative patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years of age inclusive at the time of the study who underwent colorectal surgery and are presenting for their first postoperative visit
2. Patients with a computer or phone device with video and audio capabilities

Exclusion Criteria:

1. Children <18 years of age
2. Patients with mental disability
3. Patients without a computer or phone device with video and audio capabilities
4. Patients who require physical intervention during their first postoperative visit (e.g. drain removal, suture removal, staple removal)
5. Patients who are readmitted to the hospital prior to their first postoperative visit will be excluded.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | 7 to 14 days postoperatively
  Patient satisfaction score measured by electronic survey sent to all participating patients after their first postoperative visit

SECONDARY OUTCOMES:
Patient-reported rating of safety | 7 to 14 days postoperatively
  Patient-reported sense of safety score rated from 1 to 5 with higher scores indicating greater sense of safety. This is designed to gauge how safe patients feel visiting the clinic in-person vs. online via telemedicine during the COVID pandemic
Length of visit | 7 to 14 days postoperatively
  Length of postoperative visit
Patient willingness to recommend provider to peers rated from 1 to 5 | 7 to 14 days postoperatively
  Patient willingness to recommend provider to peers rated from 1 to 5
Combined patient satisfaction score from 1st and 2nd postoperative visits | 7 to 31 days postoperatively
  Combined patient satisfaction score from 1st and 2nd postoperative visits
Distance (in kilometers) of patient's primary residence to the clinic location | 7 to 31 days postoperatively
  Distance (in kilometers) of patient's primary residence to the clinic location
60-day rate of hospital readmission | 60 days postoperatively
  Incidence of hospital readmission 60 days postoperatively
60-day rate of re-operation | 60 days postoperatively
  Incidence of re-operation 60 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Karen Zaghiyan, MD, Principal Investigator — Associate Professor of Surgery
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Grenda TR, Whang S, Evans NR 3rd. Transitioning a Surgery Practice to Telehealth During COVID-19. Ann Surg. 2020 Aug;272(2):e168-e169. doi: 10.1097/SLA.0000000000004008. PMID 32675529
- [Background] Gunter RL, Chouinard S, Fernandes-Taylor S, Wiseman JT, Clarkson S, Bennett K, Greenberg CC, Kent KC. Current Use of Telemedicine for Post-Discharge Surgical Care: A Systematic Review. J Am Coll Surg. 2016 May;222(5):915-27. doi: 10.1016/j.jamcollsurg.2016.01.062. Epub 2016 Feb 13. No abstract available. PMID 27016900
- [Background] Huang EY, Knight S, Guetter CR, Davis CH, Moller M, Slama E, Crandall M. Telemedicine and telementoring in the surgical specialties: A narrative review. Am J Surg. 2019 Oct;218(4):760-766. doi: 10.1016/j.amjsurg.2019.07.018. Epub 2019 Jul 18. PMID 31350010
- [Background] Hakim AA, Kellish AS, Atabek U, Spitz FR, Hong YK. Implications for the use of telehealth in surgical patients during the COVID-19 pandemic. Am J Surg. 2020 Jul;220(1):48-49. doi: 10.1016/j.amjsurg.2020.04.026. Epub 2020 Apr 21. PMID 32336519
- [Background] Hwa K, Wren SM. Telehealth follow-up in lieu of postoperative clinic visit for ambulatory surgery: results of a pilot program. JAMA Surg. 2013 Sep;148(9):823-7. doi: 10.1001/jamasurg.2013.2672. PMID 23842982
- [Background] Mann DM, Chen J, Chunara R, Testa PA, Nov O. COVID-19 transforms health care through telemedicine: Evidence from the field. J Am Med Inform Assoc. 2020 Jul 1;27(7):1132-1135. doi: 10.1093/jamia/ocaa072. PMID 32324855
- See also: CDC Guidelines for Healthcare Facilities — https://www.cdc.gov/coronavirus/2019-ncov/healthcare-facilities/guidance-hcf.html.
- See also: Sealed Envelope tool for randomization — https://www.sealedenvelope.com/power/binary-noninferior/